CLINICAL TRIAL: NCT04698629
Title: Pilot Study of a Community-Pharmacy Model to Expand Access to Medications to Treat and Prevent Hepatitis C, Opioid Use Disorders, Overdose and HIV Among Persons Who Inject Drugs
Brief Title: Hepatitis C Pharmacy-based Strategy for Injectors
Acronym: HepPSI
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Judith I. Tsui, Professor, School of Medicine, University of Washington
Other Study IDs: STUDY00010476; R34DA047660 (NIH)
Record Dates: First submitted 2020-11-24; First posted 2021-01-07 (Actual); Results first posted 2024-06-07 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Community Pharmacy; Direct Acting Antivirals; Patient Navigator
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is evaluate the acceptability/usage of a newly implemented model of delivery of care, namely a community-pharmacy program, to provide access to medications to treat hepatitis C (HCV), and prevent overdose and HIV, for persons who inject drugs (PWID) with HCV who are in need of treatment. Adults will be enrolled who test positive for HCV at community sites and who agree to linkage to the community-pharmacy program through the use of patient navigators. The primary outcome of the study will be the measure of the number/% of participants who are successfully linked to the community-pharmacy program and assess HCV treatment initiation, completion, and cure. In addition, other outcomes including receipt of other medications (e.g. Naloxone, pre-exposure prophylaxis (PrEP), and medications for opioid use disorders), and self-reported substance use and HIV risk behaviors will also be measured.

DETAILED DESCRIPTION:
Single-arm, prospective observational study of 40 adult persons who inject drugs (PWID) who screen positive for hepatitis C virus (HCV) with a reactive antibody test at community sites who are offered facilitated linkage to community-pharmacy program through patient navigators. Individuals who are eligible and enroll will complete a baseline survey to assess sociodemographics, substance use, HIV risk behaviors, and awareness of and interest in HCV treatment. After the survey, the participants will be linked to the community-pharmacy program, via the patient navigator, where treatment for HCV and opioid use disorder (OUD), as well as pre-exposure prophylaxis (PrEP), Naloxone and vaccinations, will be offered to participants.

After 6 months, participants will complete a follow-up survey, which will include questions on: whether an evaluation for HCV occurred at the community pharmacy, whether HCV treatment was initiated since baseline visit, substance use, HIV risk behaviors, receipt of medications to treat HCV, opioid use disorder, Naloxone and PrEP receipt, medication adherence, and injecting network.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years old
2. Reports injecting drugs with 90 days of screening
3. Positive HCV test documented (screening antibody test or viral load test)
4. Not currently taking medications to treat HCV, and never previously treated with direct-acting antivirals (DAAs) for HCV
5. Willing to undergo evaluation for HCV through a community pharmacy program and work with Patient Navigators
6. Provides release of information (ROI) to access community pharmacy program records and/or other HCV treatment providers

Exclusion Criteria:

1. People who plan to leave the Seattle area within 6 months
2. Who do not wish to be treated for their HCV infection
3. Who are known to be pregnant
4. Who report impending incarceration that would disrupt clinical care
5. Who are not comfortable reading and speaking English
6. Who report being HIV-positive
7. Who report having end-stage renal disease or require dialysis treatments
8. Who report prior enrolled in (i.e. completed at least the initial intake appointment) the Kelley-Ross pharmacy program for hepatitis C treatment ("One Step Hep C Free")

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited at various community sites in Seattle where HCV screening occurs, including syringe exchange programs, addiction treatment programs (a methadone clinic and primary care-based buprenorphine program), homeless shelters, urban drop-in shelters and low-income housing sites.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith I Tsui, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Tsui JI, Gojic AJ, Pierce KA, Tung EL, Connolly NC, Radick AC, Hunt RR, Sandvold R, Taber K, Ninburg M, Kubiniec RH, Scott JD, Hansen RN, Stekler JD, Austin EJ, Williams EC, Glick SN. Pilot study of a community pharmacist led program to treat hepatitis C virus among people who inject drugs. Drug Alcohol Depend Rep. 2023 Dec 23;10:100213. doi: 10.1016/j.dadr.2023.100213. eCollection 2024 Mar. PMID 38261893

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from community sites that serve PWID in the Seattle area: a non-profit organization with a syringe services program, an opioid treatment program, and several emergency housing units. Potential participants were identified and referred by local providers within their respective site organizations or self-referred after seeing informational flyers at study sites. The first participant was enrolled on 11/05/2020, and the last participant was enrolled on 10/28/2021.
Groups:
- Observational Group: Person who injects drugs, with documented positive hepatitis c virus test results.
Period: Overall Study
Arm/Group | Observational Group
Started | 40
Completed | 39
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Person who injects drugs, with documented positive hepatitis c virus test results.
Arm/Group | Observational Group
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (10.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Man | 24
  Woman | 12
  Non-binary or Transgender man or woman | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 6
  White | 20
  More than one race | 5
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Community Pharmacy Program Successful Linkage
Description: The number/percent of participants who successfully link to the community pharmacy program and are seen for initial evaluation.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Observational Group
Number analyzed (Participants) | 40
Participants | 38

2. Secondary Outcome: Initiation of HCV Treatment
Description: The number/percent who initiate medications for HCV.
Time Frame: 6 months
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Substance Use
Description: Compare at baseline and 6-month follow-up the number of days of drug use within the past 30 days via self-report using the modified Addition Severity Index (ASI).
Time Frame: 6 months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: HIV Drug Risk Behaviors
Description: Compare at baseline and 6-month follow-up the number of injecting episodes using shared needle/syringe within the past 30 days via self-report using the modified Risk Behaviors Survey (RBS).
Time Frame: 6 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: HIV Sex Risk Behaviors
Description: Compare at baseline and 6-month follow-up the number of episodes of unprotected vaginal or anal sex within the past 30 days via self-report using the modified Risk Behaviors Survey (RBS).
Time Frame: 6 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Utilization of Other Community Pharmacy Services
Description: The number/percent who receive of other medications (naloxone, PrEP, and medications to treat OUD) via the community pharmacy program.
Time Frame: 6 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Participant Satisfaction and Referral to the Community Pharmacy Program
Description: Self-reported participant Likert scale surveys of satisfaction and willingness to refer an injecting partner to the community pharmacy for treatment; 1=strongly disagree, 2=disagree, 3=neutral, 4=agree, 5=strongly agree with the level of satisfaction/likelihood of referral to services.
Time Frame: 6 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Completion of HCV Treatment
Description: The number/percent who complete treatment for HCV, defined as having received all planned medication doses.
Time Frame: 9 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Sustained Virologic Response (SVR12)
Description: SVR12 will be defined as undetectable HCV viral load at least 12-weeks post treatment completion.
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years
Description: Definitions for adverse event and serious adverse event used to collected adverse event information for this trial does not differ from the clinicaltrials.gov definitions. No event frequency threshold was implemented for this trial, and therefore, all events were reports
Arm/Group | Observational Group
All-Cause Mortality (participants affected / at risk) | 1/40
Serious Adverse Events (participants affected / at risk) | 2/40
Other Adverse Events (participants affected / at risk) | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observational Group (N=40)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Death (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT04698629/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/29/NCT04698629/SAP_001.pdf